CLINICAL TRIAL: NCT03362918
Title: The Impact of Continuous Aerobic Exercise and High-Intensity Interval Training on Reproductive Outcomes in Polycystic Ovary Syndrome: A Pilot Randomized Controlled Trial.
Brief Title: Polycystic Ovary Syndrome and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB17-1574
Record Dates: First submitted 2017-11-09; First posted 2017-12-05 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blind to the allocation of the study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants randomized to the control group will continue with their usual level of physical activity. They will track their menstrual cycles and perform daily ovulation tests.
  Once all post-intervention assessments are complete, they will have the option to begin an exercise program with three supervised sessions of either high-intensity interval training or continuous aerobic exercise training free of charge. They will be given a Polar heart rate (HR) monitor as a gift for their participation in the study.
- High-Intensity Interval Training (Experimental): Participants randomized to this group will complete three high intensity interval training sessions per week, two of which will be supervised. They will exercise for a total of 30 minutes per session. Each session will begin with a five-minute warm-up and end with a five-minute cool-down.
  Interventions: Behavioral: High Intensity Interval Training
- Continuous Aerobic Exercise Training (Experimental): Participants randomized to this group will complete three continuous aerobic training sessions per week, two of which will be supervised. They will exercise for a total of 50 minutes per session. Each session will begin with a five-minute warm-up and end with a five-minute cool down.
  Interventions: Behavioral: Continuous Aerobic Exercise Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — The exercise prescription is as follows:
  Type: High-Intensity Interval Training on a treadmill, elliptical trainer or cycle ergometer.
  Intensity: 30 seconds of high-intensity alternating with 90 seconds of low intensity for a total of 10 cycles
  * High intensity for most individuals will occur at approximately 90% of maximum heart rate. Using the rating of perceived exertion scale, participants should be exercising at a 9/10, which is very difficult to maintain the intensity and results in only being able to speak a few words at a time.
  * Low intensity is defined as light activity and rated as 2-3/10 on the rating of perceived exertion scale. Participants should be able to carry on a conversation and maintain the pace for hours.
  Duration: 30 minutes Frequency: 3 times per week
  Arms: High-Intensity Interval Training
Behavioral: Continuous Aerobic Exercise Training — The exercise prescription for the continuous aerobic exercise group is as follows:
  Type: Aerobic exercise including walking, running, cycling or using the elliptical trainer.
  Intensity: Moderate intensity, defined as 50-60% of the participant's maximum heart rate. On the rating of perceived exertion scale, this corresponds with a 4-6/10, which allows participants to hold a conversation while breathing heavily.
  Duration: 50 minutes Frequency: 3 times per week
  Arms: Continuous Aerobic Exercise Training

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a common hormonal disorder characterized by oligo-ovulatory menstrual dysfunction, androgen excess and polycystic ovaries. It affects ten to fifteen percent of reproductive-age women and has been associated with complications in reproductive, metabolic and cardiovascular health. Current Clinical Practice Guidelines suggest exercise and weight loss for PCOS, although their specific roles in improving PCOS-related symptoms are uncertain.

Non-pharmacological treatments are appealing to many reproductive age women. There is preliminary evidence that exercise in PCOS may increase menstrual regularity, ovulation, cardiorespiratory fitness, health-related quality of life (HRQOL) and self-esteem, and decrease body fat and insulin resistance. These studies have been limited by short durations and lack of randomization or appropriate control groups.

High-intensity interval training (HIIT), which involves brief intervals of near-maximal exercise alternating with lower-intensity exercise, is becoming increasingly popular in the exercise community. In some non-PCOS trials, HIIT resulted in improved cardiovascular fitness and greater fat loss compared with continuous aerobic exercise. No other trials are currently on-going that are comparing HIIT with continuous aerobic exercise training in women with PCOS (as confirmed by searches of the literature and the clinical trials registry maintained by the US NIH).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for inclusion if they are females between the ages of 18 and 40 years with a diagnosis of PCOS according to the 2003 revised Rotterdam criteria, confirmed by a qualified member of our research team. Participants will have at least two of the three following criteria:

  1. Oligo-ovulation or anovulation. Oligo-ovulation is defined as menstrual cycles greater than 35 days or less than 8 menstrual cycles per year. Anovulation is defined as no ovulation in more than 90 days.
  2. Clinical and/or biochemical signs of hyperandrogenism. Clinical hyperandrogenism is defined as a modified Ferriman Gallwey score greater than or equal to 8. Biochemical hyperandrogenism is defined as a free androgen index greater than or equal to 5.1.
  3. Polycystic ovaries defined as the presence of 12 or more follicles in each ovary measuring 2-9 mm in diameter, and/or increased ovarian volume (>10 mL).

Exclusion Criteria:

* Participants must not have a diagnosis of or clinical evidence of Cushing's syndrome, androgen-secreting tumours, congenital adrenal hyperplasia including classical and non-classical, uncontrolled thyroid dysfunction, diabetes, hemoglobin A1c greater than or equal to 6.5%, hypogonadotropic hypogonadism, premature ovarian insufficiency, or hyperprolactinemia.
* Participants must not be pregnant or breastfeeding within the three months prior to enrolment and must not be using or have used a hormonal contraceptive within three months of enrolment.
* Participants will be excluded if they are taking any medications to treat insulin resistance including metformin, medications likely to increase insulin resistance such as corticosteroids, or any medications that may affect ovulation including clomiphene citrate, letrozole, or gonadotropins. They must not be taking medications to treat hirsutism including spironolactone.
* Participants must not be habitually exercising more than two times per week for more than twenty minutes per session.
* Participants must be able to participate in the exercise intervention, therefore will be excluded if they have a physical injury, illness or disability that prevents them from doing so.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Ovulation Rate | Up to 9 months.
  The ovulation rate is defined as the number of times a participant ovulates during the intervention period adjusted for the baseline ovulation rate during the run-in phase.

SECONDARY OUTCOMES:
Hirsutism | Up to 9 months.
  This will be assessed using the Ferriman-Gallwey Score, which quantifies hair growth in women with PCOS. Scores range from 0-36, with higher scores indicating more hair growth.
Menstrual Cycle Length | Up to 9 months.
  The menstrual cycle starts on the first day of menses and lasts until menses resumes. A regular menstrual cycle length ranges from 24 to 35 days.
Luteal Phase Length | Up to 9 months.
  The luteal phase length is defined as the number of days from ovulation to menses (normal is 12 to 16 days).
Pregnancy | Up to 15 months.
  Pregnancy will be confirmed by the presence of a fetal heart beat on a first-trimester ultrasound, ordered by the participant's physician.
Spontaneous Abortions | Up to 15 months.
  Non-induced embryonic or fetal death or passage of products of conception before 20 weeks gestation.
Live Births | Up to 15 months.
  The delivery of a live infant
Body Weight | Up to 9 months.
  Change in body weight pre- and post-intervention
Body Mass Index | Up to 9 months.
  Change in body mass index pre- and post-intervention
Waist Circumference | Up to 9 months.
  Change in waist circumference pre- and post-intervention
Blood Pressure | Up to 9 months.
  Change in blood pressure pre- and post-intervention
Hemoglobin A1c | Up to 9 months.
  Change in hemoglobin A1c pre- and post-intervention
Fasting Glucose | Up to 9 months.
  Change in fasting glucose pre- and post-intervention
Fasting Insulin | Up to 9 months.
  Change in fasting insulin pre- and post-intervention
Homeostatic Model of Insulin Resistance (HOMA-IR) | Up to 9 months.
  Change in HOMA-IR pre- and post-intervention
HOMA-2 | Up to 9 months.
  To assess insulin resistance using the updated HOMA-2 model
Lipids - total cholesterol, LDL, HDL, triglycerides | Up to 9 months.
  Change in lipid profile pre- and post-intervention
Liver Enzymes - ALT, GGT | Up to 9 months.
  Change in liver enzymes pre- and post-intervention
Cardiorespiratory Fitness | Up to 9 months.
  Change in cardiorespiratory fitness assessed as maximal oxygen consumption evaluated using a treadmill test and a metabolic cart
Health-Related Quality of Life | Up to 15 months.
  Change in Health-Related Quality of Life using the PCOS-Q and SF-36
Obstructive Sleep Apnea | Up to 9 months.
  Change in symptoms of obstructive sleep apnea pre- and post-intervention using the STOP-BANG score. This score has 8 questions, and the likelihood of obstructive sleep apnea increases with a score of 3 or more.
Participant Satisfaction | Up to 9 months.
  To assess participant satisfaction with their participation in this study using a questionnaire specifically designed for this study, with higher numbers indicating higher satisfaction.
Participant Recruitment - Number of Participants Screened | Up to enrolment in study.
  Participant recruitment will be assessed by recording the number of participants that were initially screened.
Participant Recruitment - Recruitment Method | Up to enrolment in study.
  The investigators will document how each participant was recruited (i.e. poster, physician referral, etc.).
Participant Recruitment - Number of Participants That Met Criteria | Up to enrolment in the study.
  The investigators will record the number that met all inclusion and exclusion criteria.
Participant Recruitment - Number of Participants That Signed Informed Consent | Up to enrolment in the study.
  The investigators will record the number that agreed to participate in the study and signed informed consent.
Participant Dropout | Up to 15 months.
  Dropout will be reported as a percentage of participants that enrolled in the study and did not complete the study.
Adherence to Menstrual Cycle Tracking | Up to 9 months.
  Participants will record features of their menstrual cycle daily (menses, spotting, no menstrual bleeding) using a monthly calendar, or phone app. Adherence will be recorded as the percentage of data recorded over the study duration.
Adherence to Ovulation Prediction Kit (OPK) Testing | Up to 9 months.
  Participants will complete the OPK test daily, take a digital photograph of the used test strip and send it to the research team daily. Adherence will be recorded as the percentage completed over the study.
Adherence to Exercise Sessions | Up to 9 months.
  For individuals randomized to the high-intensity training group or the continuous aerobic exercise training group, exercise sessions will be tracked using a Polar heart rate monitor and data will be downloaded weekly at a supervised exercise session. Participants will also log their workouts (type, duration, intensity) in a log book.
Change in Gut Microbiota Composition | Up to 9 months.
  Pre- and post-intervention stool samples will be assessed with 16S rRNA sequencing.
Daily Physical Activity Level | Up to 9 months.
  All individuals will wear Polar A370 fitness trackers during the intervention phase, and daily steps and kilocalories per day will be recorded.
Physical Activity Enjoyment | Up to 9 months.
  Individuals randomized to the exercise groups will complete the Physical Activity Enjoyment Scale during an exercise training session at the beginning of the exercise intervention, at 3 months into the intervention and at 6 months into the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Sigal, MD, MPH, Principal Investigator — University of Calgary, rsigal@ucalgary.ca
Locations (1):
- University of Calgary Clinical Trials Unit, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lizneva D, Suturina L, Walker W, Brakta S, Gavrilova-Jordan L, Azziz R. Criteria, prevalence, and phenotypes of polycystic ovary syndrome. Fertil Steril. 2016 Jul;106(1):6-15. doi: 10.1016/j.fertnstert.2016.05.003. Epub 2016 May 24. PMID 27233760
- [Background] Sirmans SM, Pate KA. Epidemiology, diagnosis, and management of polycystic ovary syndrome. Clin Epidemiol. 2013 Dec 18;6:1-13. doi: 10.2147/CLEP.S37559. PMID 24379699
- [Background] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499
- [Background] Legro RS, Arslanian SA, Ehrmann DA, Hoeger KM, Murad MH, Pasquali R, Welt CK; Endocrine Society. Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2013 Dec;98(12):4565-92. doi: 10.1210/jc.2013-2350. Epub 2013 Oct 22. PMID 24151290
- [Background] Thomson RL, Buckley JD, Noakes M, Clifton PM, Norman RJ, Brinkworth GD. The effect of a hypocaloric diet with and without exercise training on body composition, cardiometabolic risk profile, and reproductive function in overweight and obese women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Sep;93(9):3373-80. doi: 10.1210/jc.2008-0751. Epub 2008 Jun 26. PMID 18583464
- [Background] Turan V, Mutlu EK, Solmaz U, Ekin A, Tosun O, Tosun G, Mat E, Gezer C, Malkoc M. Benefits of short-term structured exercise in non-overweight women with polycystic ovary syndrome: a prospective randomized controlled study. J Phys Ther Sci. 2015 Jul;27(7):2293-7. doi: 10.1589/jpts.27.2293. Epub 2015 Jul 22. PMID 26311969
- [Background] Vizza L, Smith CA, Swaraj S, Agho K, Cheema BS. The feasibility of progressive resistance training in women with polycystic ovary syndrome: a pilot randomized controlled trial. BMC Sports Sci Med Rehabil. 2016 May 11;8:14. doi: 10.1186/s13102-016-0039-8. eCollection 2016. PMID 27175282
- [Background] Aubuchon M, Laughbaum N, Poetker A, Williams D, Thomas M. Supervised short-term nutrition and exercise promotes weight loss in overweight and obese patients with polycystic ovary syndrome. Fertil Steril. 2009 Apr;91(4 Suppl):1336-8. doi: 10.1016/j.fertnstert.2008.03.028. Epub 2008 Jun 13. PMID 18555225
- [Background] Nybacka A, Carlstrom K, Stahle A, Nyren S, Hellstrom PM, Hirschberg AL. Randomized comparison of the influence of dietary management and/or physical exercise on ovarian function and metabolic parameters in overweight women with polycystic ovary syndrome. Fertil Steril. 2011 Dec;96(6):1508-13. doi: 10.1016/j.fertnstert.2011.09.006. Epub 2011 Sep 29. PMID 21962963
- [Background] Jedel E, Labrie F, Oden A, Holm G, Nilsson L, Janson PO, Lind AK, Ohlsson C, Stener-Victorin E. Impact of electro-acupuncture and physical exercise on hyperandrogenism and oligo/amenorrhea in women with polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E37-45. doi: 10.1152/ajpendo.00495.2010. Epub 2010 Oct 13. PMID 20943753
- [Background] Thomson RL, Buckley JD, Brinkworth GD. Exercise for the treatment and management of overweight women with polycystic ovary syndrome: a review of the literature. Obes Rev. 2011 May;12(5):e202-10. doi: 10.1111/j.1467-789X.2010.00758.x. PMID 20546140
- [Background] Batacan RB Jr, Duncan MJ, Dalbo VJ, Tucker PS, Fenning AS. Effects of high-intensity interval training on cardiometabolic health: a systematic review and meta-analysis of intervention studies. Br J Sports Med. 2017 Mar;51(6):494-503. doi: 10.1136/bjsports-2015-095841. Epub 2016 Oct 20. PMID 27797726
- [Derived] Benham JL, Booth JE, Friedenreich CM, Rabi DM, Sigal RJ. Comparative Success of Recruitment Strategies for an Exercise Intervention Trial Among Women With Polycystic Ovary Syndrome: Observational Study. J Med Internet Res. 2021 Mar 30;23(3):e25208. doi: 10.2196/25208. PMID 33783363